CLINICAL TRIAL: NCT00486824
Title: Indocin Versus Nifedipine for Preterm Labor Tocolysis - A Randomized Double-Blinded Clinical Trial
Brief Title: Indomethacin Versus Nifedipine for Preterm Labor Tocolysis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Deirdre Judith Lyell, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 97873
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-08

CONDITIONS: Obstetric Labor, Premature
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Indomethacin; Nifedipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indomethacin (Active Comparator): 50 mg. oral Indomethacin initially, followed by 25 mg every 6 hrs for 48 hrs.
  Interventions: Drug: Indomethacin
- Nifedipine (Active Comparator): 30 mg Nifedipine initially followed by 20 mg every 6 hrs for 48 hrs.
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Indomethacin — One 50 mg tablet of Indomethacin plus 2 pills of placebo followed by one 25 mg tablet of oral indomethacin every 6 hrs for 48 hrs.
  Arms: Indomethacin
Drug: Nifedipine — Three 10 mg tablets of Nifedipine followed by one 20 mg tablet every 6 hrs for 48 hrs.
  Arms: Nifedipine

SUMMARY:
Indomethacin and Nifedipine are commonly used medications for treatment of pre term labor. This study will compare the efficacy and adverse outcomes of oral nifedipine versus oral indomethacin for preterm labor tocolysis in an effort to identify which drug is most effective.

Patients diagnosed with preterm labor who grant consent will be randomized by the pharmacy to receive oral nifedipine or oral indomethacin. Both the patient and primary medical provider will be blinded to the identity of the study drug. An abdominal ultrasound will be performed in the labor and delivery unit prior to the administration of the tocolytic in order to assess fetal position and fluid level, and to document fetal cardiac activity and movement, and will be repeated at 48 hours post-randomization. Following randomization, the patient will be given either 50 mg oral indomethacin with two pills of placebo, or 3 pills each containing 10 mg oral nifedipine for a total of 30 mg. The patients will then receive either 25 mg of oral indomethacin every 6 hours for 48 hours, or 20 mg of oral nifedipine every 6 hours for 48 hours. Tocolysis beyond 48 hours will not be used.

DETAILED DESCRIPTION:
Patients presenting between 24-34 weeks gestation diagnosed with preterm labor who grant consent will be randomized by the pharmacy to receive oral nifedipine or oral indomethacin. Both the patient and primary medical provider will be blinded to the identity of the study drug. An abdominal ultrasound will be performed in the labor and delivery unit prior to the administration of the tocolytic in order to assess fetal position and fluid level, and to document fetal cardiac activity and movement, and will be repeated at 48 hours post-randomization. Following randomization, the patient will be given either 50 mg oral indomethacin with two pills of placebo, or 3 pills each containing 10 mg oral nifedipine for a total of 30 mg. The patients will then receive either 25 mg of oral indomethacin every 6 hours for 48 hours, or 20 mg of oral nifedipine every 6 hours for 48 hours. Tocolysis beyond 48 hours will not be used. Antibiotics and steroids for fetal lung maturity will be administered as per standard of care for preterm labor. Maternal side effects and delivery outcomes will be assessed from questionnaires administered by the study team following treatment, and/or from review of the patient's medical records.

ELIGIBILITY:
Inclusion Criteria:

* Singleton and twin gestations
* Intact amniotic membranes
* No contra-indications to tocolysis
* 24-34 weeks gestation by last menstrual period and/or ultrasound
* Documented cervical change, and regular painful uterine contractions at least every 5 minutes, or at least 2 cm cervical dilation and 80% effacement

Exclusion Criteria:

* Ruptured amniotic membranes
* Signs/symptoms of chorioamnionitis (maternal temperature greater than 100.4 F/38.0 C, fetal tachycardia, uterine tenderness)
* Non-reassuring fetal heart rate tracings
* Contra-indications to indomethacin or nifedipine
* Contra-indications to tocolysis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2012-12-08 (Actual); Study Completion 2012-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Judith Lyell, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 29 patients were initially consented and enrolled. Patients were enrolled through December 2012 but protocol remained open until 2018. Due to patient privacy regulations, the data were accessible for only 10 patients.
Groups:
- Nifedipine: 30 mg Nifedipine initially followed by 10 mg every 6 hrs for 48 hrs.
  Nifedipine: Three 10 mg tablets of Nifedipine followed by one 20 mg tablet every 6 hrs for 48 hrs.
Period: Overall Study
Arm/Group | Indomethacin | Nifedipine
Started | 5 | 5
Completed | 3 | 3
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: Data were accessible for limited participants due to patient privacy regulations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Indomethacin | Nifedipine | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 26.0 [20.0 to 37.0] | 30 [19.0 to 37.0] | 26.5 [19.0 to 37.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Count of Patients With Recurrent Preterm Labor Within Two Weeks of Randomization
Description: Preterm labor was defined as documented cervical change and regular uterine contractions at least every 5 minutes, or at least 2 cm cervical dilation and 80% cervical effacement. Preterm labor is defined as uterine contractions occurring up to 37 weeks of pregnancy.
Time Frame: Two weeks after enrolled and randomized, up to 37 weeks of pregnancy
Population: Participants with accessible data are included in the analysis. Not all data were accessible due to patient data privacy regulations.
Measure: Count of Participants; unit: Participants
Arm/Group | Indomethacin | Nifedipine
Number analyzed (Participants) | 5 | 5
Participants | 2 | 1
Statistical Analysis 1: Comparison: Indomethacin vs Nifedipine; Test type: Superiority; p = 0.004, Fisher Exact

2. Secondary Outcome: Neonatal Birthweight
Description: Birthweight is presented in grams
Time Frame: Until discharge of mother and neonate from delivery hospital, up to 30 days after delivery
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Indomethacin | Nifedipine
Number analyzed (Participants) | 5 | 5
grams | 2830 [2750 to 2880] | 2240 [2000 to 2740]

3. Secondary Outcome: Gestational Age at Delivery
Time Frame: Up to 42 weeks of pregnancy
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Indomethacin | Nifedipine
Number analyzed (Participants) | 5 | 5
weeks | 37.0 [35.0 to 37.4] | 34.0 [33.4 to 38.0]

4. Secondary Outcome: Days From First Medication Initiation to Delivery as a Measure of Delay in Delivery
Time Frame: Up to 42 weeks of pregnancy
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Indomethacin | Nifedipine
Number analyzed (Participants) | 5 | 5
days | 34.0 [22.0 to 77.0] | 36.0 [28.0 to 52.0]

5. Secondary Outcome: Count of Participants With Neonatal Morbidity
Description: Neonatal morbidity included admission to neonatal intensive care unit, respiratory distress or sepsis.
Time Frame: Up to 42 weeks of pregnancy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Indomethacin | Nifedipine
Number analyzed (Participants) | 5 | 5
Participants | 2 | 3

6. Secondary Outcome: Count of Participants With Side-effect Due to the Medication
Description: Monitored side-effects for this outcome included abdominal pain, blood pressure change, GI-symptoms and skin rash.
Time Frame: Up to 42 weeks of pregnancy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Indomethacin | Nifedipine
Number analyzed (Participants) | 5 | 5
Participants | 2 | 3

7. Secondary Outcome: Time to Uterine Quiescence
Description: Uterine quiescence was defined as six or fewer uterine contractions per hour. Outcome was described as days.
Time Frame: Up to 42 weeks of pregnancy
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Indomethacin | Nifedipine
Number analyzed (Participants) | 5 | 4
days | 2.0 [2.0 to 4.0] | 2.0 [1.75 to 2.25]

ADVERSE EVENTS:
Time Frame: Up to maternal and neonatal discharge from the delivery hospital, up to 30 days after the delivery.
Arm/Group | Indomethacin | Nifedipine
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indomethacin (N=5) | Nifedipine (N=5)
Gastrointestinal symptoms (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hypotension (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The sample size for the analysis was not reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes